CLINICAL TRIAL: NCT06883344
Title: Automated Insulin for Management of Intrapartum Glycemia (AIMING): a Randomized Clinical Trial
Brief Title: Automated Insulin for Management of Intrapartum Glycemia
Acronym: AIMING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-43619
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes (T1D); Pregnancy; Pre-Gestational Diabetes
Keywords: Pregnancy; Intrapartum glycemic management; Neonatal hypoglycemia; Perinatal care; Diabetes in pregnancy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes, Gestational | interventions — Insemination, Artificial, Heterologous; Drug Delivery Systems; Insulin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intravenous (IV) insulin (Active Comparator)
  Interventions: Other: Intravenous (IV) insulin
- Automated insulin delivery (AID) system (Experimental)
  Interventions: Device: Automated insulin delivery (AID) system

INTERVENTIONS:
Device: Automated insulin delivery (AID) system — An AID system incorporates data from a continuous glucose monitor (CGM) to automatically adjust the amount of insulin delivered by an insulin pump via an algorithm that incorporates multiple factors, including predicted glucose level in the next 30-60 minutes, target glucose level, and recent insulin delivery.
  Arms: Automated insulin delivery (AID) system
Other: Intravenous (IV) insulin — Variable rate IV insulin infusions are used in most labor/delivery units as the standard of care for glycemic management for pregnant people with T1D. A continuous rate of IV insulin is infused, with manual rate adjustments made based on current glucose level and hospital-specific protocols.
  Arms: Intravenous (IV) insulin

SUMMARY:
The goal of this clinical trial is learn if automated insulin delivery (AID) systems can be used for glucose management during labor/delivery for pregnant people with type 1 diabetes (T1D). The main questions this study aims to answer are

* What are the neonatal glycemic outcomes with use of AID systems during labor/delivery?
* Do patients report higher birth satisfaction with use of AID systems during labor/delivery?
* Are glycemic parameters like time-in-range (TIR) better with use of AID systems during labor/delivery?

Researchers will compare AID systems to intravenous (IV) insulin (the current standard of care for glucose management during labor/delivery) by randomly assigning participants to one or the other.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant at ≥ 34 weeks
* Known diagnosis of type 1 diabetes ≥ 1 year
* Use of commercially available AID system since at least 28 weeks gestation
* Singleton pregnancy
* English- or Spanish-speaking

Exclusion Criteria:

* Multifetal gestation
* Planned cesarean delivery
* Use of medications known to interfere with glucose metabolism
* Intrauterine fetal demise
* Physical or psychological disease likely to interfere with the conduct of the study and/or the ability to participate in own healthcare

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
First neonatal glucose value | Within 2 hours of birth
  A primary clinical goal of intrapartum glycemic management is to minimize the likelihood of low neonatal glucose values (hypoglycemia).

SECONDARY OUTCOMES:
Birth Satisfaction Scale Revised (BSS-R) score | Within 2 weeks of delivery
  The BSS-R is a 10-item, multi-dimensional, psychometric instrument that has been validated as a measure of birth satisfaction. This endpoint was selected to adequately assess patient perception of quality of care received and labor-related stress experienced.
CGM-derived glycemic parameters | From admission to labor/delivery unit to birth of infant
  Glycemic parameters like time in range (TIR), time below range (TBR), and time above range (TAR) will be examined as markers of intrapartum glycemia

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Sobhani, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes